CLINICAL TRIAL: NCT01435187
Title: Prematurity and Respiratory Outcomes Program (PROP) Core Database Protocol
Brief Title: Prematurity and Respiratory Outcomes Program (PROP)
Acronym: PROP
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 813839; U01HL101794-02 (NIH)
Record Dates: First submitted 2011-09-14; First posted 2011-09-16 (Estimated); Last update posted 2016-11-07 (Estimated); Status verified 2016-11

CONDITIONS: Prematurity; Respiratory Disease
MeSH Terms: conditions — Premature Birth; Respiration Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva for DNA, Urine and Tracheal Aspirate
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Infant Pulmonary Function Testing (iPFT): A standardized method of performing infant PFTs using the raised volume rapid thoracoabdominal compression (RVRTC) technique will be used. This test will be performed on infants at one year (corrected age). The target sample size of 180 studies will represent the largest number of RVRTC PFTs in the preterm population and will enhance study of the relationship between lung function at 1 year of age and clinical and biologic factors associated with respiratory disease. Although the primary PFT measures will be derived from RVRTC, V'maxFRC, respiratory system compliance (Crs) and resistance (Rrs) will also be measured because these can be easily obtained. Crs and Rrs will be obtained using the single breath occlusion method.

SUMMARY:
In survivors of extreme prematurity to 36 weeks Post Menstrual Age (PMA), specific biologic, physiologic and clinical data obtained during the initial hospitalization will predict respiratory morbidity as defined by respiratory health care utilization and respiratory symptoms, between discharge and 1 year corrected age.

This protocol describes a collaboratively developed multicenter study of very preterm infants from birth through the time of discharge from the Neonatal Intensive Care Unit (NICU) and up to 1 year of age, corrected for the degree of prematurity.

DETAILED DESCRIPTION:
The primary goal of the PROP studies is to identify biomarkers (biochemical, physiological and genetic) and clinical variables that are associated with and thus potentially predictive of pulmonary status in preterm infants up to 1 year corrected age. An objective and validated measure of pulmonary outcome at 1 year does not currently exist. Some promising measures are in development but not yet ready for use in a multi-center large clinical study.

Moreover, the burden of chronic respiratory illness on the infants and their families is of utmost importance. A composite primary outcome of morbidity that is based on serial parental reports of respiratory symptoms, medications, hospitalizations and dependence on technology during the first year of life has been developed.

Data collection for the outcome assessment will be based on interviews conducted with the infant's main caregiver at 3, 6, 9 and 12 months corrected age. The time frame for data collection is based on questions "since last contact." Numerous epidemiological studies of asthma have used parental or self report of symptoms, physician-diagnosed asthma and allergies, or the use of medications (which may abrogate symptoms) as critical outcomes.

Survey items selected for the determination of the primary outcome will be focused on the following four domains, with any positive response to any element identifying morbidity:

1. Respiratory medications: inhaled bronchodilators, inhaled steroids, systemic steroids, methylxanthines, diuretics, pulmonary vasodilators
2. Hospitalizations for cardiopulmonary causes: any hospitalization regardless of duration
3. Symptoms: any wheeze, cough without cold
4. Home technology dependence: use of home oxygen, ventilator or continuous positive airway pressure (CPAP or BiPAP) of any duration since last contact

The primary outcome will be dichotomous, and defined as "No substantial post-prematurity respiratory disease" or "Post-prematurity respiratory disease." To be classified as having post-prematurity respiratory disease, infants must have a positive response in at least 1 of 4 morbidity domains during at least 2 separate parental interviews. Quarterly data collection up to 1 year corrected age will allow us to identify phenotypes based on the trajectory of post-prematurity respiratory disease and how these different trajectories predict later lung function and the diagnosis of asthma, if we continue to follow this cohort of children.

During hospitalization, all centers will obtain samples of tracheal aspirate, urine and saliva (for DNA extraction) from enrolled infants. At 36 weeks PMA, infants will have respiratory assessments dependent upon their respiratory status: i) respiratory inductive plethysmography (RIP) assesses alterations in tidal breathing resulting from reduced lung compliance and airway obstruction, ii) and a room air challenge (RAC).

ELIGIBILITY:
Inclusion Criteria:

* Infants who are less than or equal to 7 days old
* Gestational Age (GA) between 23 weeks and 0/7 days and 28 weeks and 6/7 days

Exclusion Criteria:

* Infants who meet any of the following conditions will be excluded from the PROP cohort:

  1. The infant is not considered to be viable (decision made not to provide life-saving therapies)
  2. Congenital heart disease (not including PDA and hemodynamically insignificant VSD or ASD)
  3. Structural abnormalities of the upper airway, lungs or chest wall
  4. Other congenital malformations or syndromes that adversely affect life expectancy or cardio-pulmonary development
  5. Family is unlikely to be available for long-term follow-up

Ages: 1 Day to 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants admitted to the Neonatal Intensive Care Unit who are < 29 weeks gestational age
Sampling Method: Non-Probability Sample
Enrollment: 835 (Actual)
Dates: Start 2011-08; Primary Completion 2015-04 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Respiratory morbidity | 1 year (corrected age)
  The primary goal of the PROP studies (single center and multicenter protocols) is to identify biomarkers (biochemical, physiological and genetic) and clinical variables that are associated with and thus potentially predictive of pulmonary status in preterm infants up to 1 year corrected age.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara K Schmidt, MD, Principal Investigator — University of Pennsylvania; Jonas H Ellenberg, PhD, Principal Investigator — University of Pennsylvania; Gloria S Pryhuber, MD, Principal Investigator — University of Rochester; Alan H Jobe, MD, PhD, Principal Investigator — Cincinnati Childrens Hospital; Aaron Hamvas, MD, Principal Investigator — Washington University School of Medicine / St. Louis Children's Hospital; Judy Aschner, MD, Principal Investigator — Vanderbilt University School of Medicine; Roberta L Keller, MD, Principal Investigator — University of California San Francisco/Benioff Children's Hospital; Judith Voynow, MD, Principal Investigator — Duke University; Stephanie D Davis, MD, Principal Investigator — Indiana University/Riley Hospital for Children
Locations (13):
- United States (13):
  - Alta Bates Summit Medical Center, Oakland, California
  - University of California, San Francisco, San Francisco, California
  - Indiana University Health/Riley Hospital for Children, Indianapolis, Indiana
  - Washington Universitiy, St Louis, Missouri
  - University of Buffalo, Buffalo, New York
  - University of Rochester, Rochester, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati University Hospital, Cincinnati, Ohio
  - Good Samaritan Hospital, Cincinnati, Ohio
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Jackson-Madison County General Hospital, Jackson, Tennessee
  - Monroe Carell Jr Children's Hospital at Vanderbilt, Nashville, Tennessee
  - University of Texas, Houston, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Maitre NL, Ballard RA, Ellenberg JH, Davis SD, Greenberg JM, Hamvas A, Pryhuber GS; Prematurity and Respiratory Outcomes Program. Respiratory consequences of prematurity: evolution of a diagnosis and development of a comprehensive approach. J Perinatol. 2015 May;35(5):313-321. doi: 10.1038/jp.2015.19. Epub 2015 Mar 26. PMID 25811285
- [Background] Pryhuber GS, Maitre NL, Ballard RA, Cifelli D, Davis SD, Ellenberg JH, Greenberg JM, Kemp J, Mariani TJ, Panitch H, Ren C, Shaw P, Taussig LM, Hamvas A; Prematurity and Respiratory Outcomes Program Investigators. Prematurity and respiratory outcomes program (PROP): study protocol of a prospective multicenter study of respiratory outcomes of preterm infants in the United States. BMC Pediatr. 2015 Apr 10;15:37. doi: 10.1186/s12887-015-0346-3. PMID 25886363
- [Background] Poindexter BB, Feng R, Schmidt B, Aschner JL, Ballard RA, Hamvas A, Reynolds AM, Shaw PA, Jobe AH; Prematurity and Respiratory Outcomes Program. Comparisons and Limitations of Current Definitions of Bronchopulmonary Dysplasia for the Prematurity and Respiratory Outcomes Program. Ann Am Thorac Soc. 2015 Dec;12(12):1822-30. doi: 10.1513/AnnalsATS.201504-218OC. PMID 26397992
- [Derived] Dylag AM, Kopin HG, O'Reilly MA, Wang H, Davis SD, Ren CL, Pryhuber GS. Early Neonatal Oxygen Exposure Predicts Pulmonary Morbidity and Functional Deficits at 1 Year. J Pediatr. 2020 Aug;223:20-28.e2. doi: 10.1016/j.jpeds.2020.04.042. PMID 32711747
- [Derived] Voynow JA, Fisher K, Sunday ME, Cotten CM, Hamvas A, Hendricks-Munoz KD, Poindexter BB, Pryhuber GS, Ren CL, Ryan RM, Sharp JK, Young SP, Zhang H, Greenberg RG, Herring AH, Davis SD. Urine gastrin-releasing peptide in the first week correlates with bronchopulmonary dysplasia and post-prematurity respiratory disease. Pediatr Pulmonol. 2020 Apr;55(4):899-908. doi: 10.1002/ppul.24665. Epub 2020 Jan 29. PMID 31995668
- [Derived] Ren CL, Feng R, Davis SD, Eichenwald E, Jobe A, Moore PE, Panitch HB, Sharp JK, Kisling J, Clem C, Kemp JS. Tidal Breathing Measurements at Discharge and Clinical Outcomes in Extremely Low Gestational Age Neonates. Ann Am Thorac Soc. 2018 Nov;15(11):1311-1319. doi: 10.1513/AnnalsATS.201802-112OC. PMID 30088802
- [Derived] Blaisdell CJ, Troendle J, Zajicek A; Prematurity and Respiratory Outcomes Program. Acute Responses to Diuretic Therapy in Extremely Low Gestational Age Newborns: Results from the Prematurity and Respiratory Outcomes Program Cohort Study. J Pediatr. 2018 Jun;197:42-47.e1. doi: 10.1016/j.jpeds.2018.01.066. Epub 2018 Mar 26. PMID 29599068
- [Derived] Keller RL, Feng R, DeMauro SB, Ferkol T, Hardie W, Rogers EE, Stevens TP, Voynow JA, Bellamy SL, Shaw PA, Moore PE; Prematurity and Respiratory Outcomes Program. Bronchopulmonary Dysplasia and Perinatal Characteristics Predict 1-Year Respiratory Outcomes in Newborns Born at Extremely Low Gestational Age: A Prospective Cohort Study. J Pediatr. 2017 Aug;187:89-97.e3. doi: 10.1016/j.jpeds.2017.04.026. Epub 2017 May 17. PMID 28528221